CLINICAL TRIAL: NCT01715870
Title: Life Style and Food Habits Questionnaire in the Portuguese Population Aged 55 or More.
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Principal Investigator, Rufino Silva, MD, PhD, Association for Innovation and Biomedical Research on Light and Image
Other Study IDs: 4C-2012-04
Record Dates: First submitted 2012-10-23; First posted 2012-10-29 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Age Related Macular Degeneration
Keywords: Age related macular degeneration; Food habits; Life style; Risk factors; questionnaire
MeSH Terms: conditions — Macular Degeneration; Feeding Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Population of the "Epidemiological study on AMD".
  Interventions: Behavioral: Life style and food habits questionnaire

INTERVENTIONS:
Behavioral: Life style and food habits questionnaire

SUMMARY:
The study population will be selected from the "Epidemiological study on the prevalence of Age related Macular Degeneration in Portugal" (Protocol N. CC-01-2009) where retinal photographic grading (current gold standard for AMD assessment) was performed to confirm AMD diagnostic. This study provides a population-based sample in which precise and contemporary information on the frequency of nutritional and lifestyle risk factors will be collected, enabling to evaluate whether the separate and/or joint effects of these factors, if found significant, are likely to have a major public health impact in terms of AMD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in the Epidemiologic Study (Protocol N. CC-01-2009). (Subjects aged over 55 years-old included in health care units of Mira or Lousã).
* Written Informed Consent Form signed.

Exclusion Criteria:

- None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects that participated in the "Epidemiological study on the prevalence of Age related Macular Degeneration in Portugal" (Protocol N. CC-01-2009) will be invited to answer a validated life style and food habits questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Life style and food habits questionnaire. | 2 years
  Life style and food habits questionnaire. (This questionnaire assesses life style habits such as physical exercise and smoking habits and quantifies dietary intake.)

CONTACTS AND LOCATIONS:
Overall Officials: Rufino M Silva, MD, PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Derived] Barreto P, Farinha C, Coimbra R, Cachulo ML, Melo JB, Lechanteur Y, Hoyng CB, Cunha-Vaz J, Silva R. Interaction between genetics and the adherence to the Mediterranean diet: the risk for age-related macular degeneration. Coimbra Eye Study Report 8. Eye Vis (Lond). 2023 Aug 14;10(1):38. doi: 10.1186/s40662-023-00355-0. PMID 37580831